CLINICAL TRIAL: NCT05283031
Title: The Water Drinking Test in Glaucoma Study
Acronym: WIGS
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 19IC5525
Record Dates: First submitted 2022-03-07; First posted 2022-03-16 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: Glaucoma
Keywords: Intraocular Pressure; Stress Test; Correlation; Water Drinking Test; OCT; Normal Tension Glaucoma
MeSH Terms: conditions — Glaucoma; Low Tension Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Modified Diurnal Tension Curve — The modified diurnal tension curve (mDTC), an alternative that involves IOP measurements every 2 or 3 hours during office hours, is more feasible and may provide better information regarding the IOP profile than single IOP measurements.

SUMMARY:
To investigate the correlation and agreement between the intraocular pressure peaks detected during the water drinking test and modified diurnal tension curve in glaucomatous eyes and to analyse whether this is associated with prognostic outcome. The study will also measure autonomic nervous system activation during the test to investigate one possible mechanism behind it.

DETAILED DESCRIPTION:
Glaucoma is a progressive optic neuropathy characterized by progressive loss of retinal ganglion cells, leading to thinning of the retinal nerve fiber layer and visual field losses. It is the leading cause of irreversible blindness in the world [2] and affects more than 70 million people worldwide. Intraocular pressure (IOP) is the main risk factor for the development and progression of glaucoma. The gold standard for intraocular pressure (IOP) measurement is applanation tonometry. Routine office measurements may not detect IOP peaks in roughly 30% of patients due to variation throughout the day and this detection failure may be responsible for visual field progression in apparently well-controlled patients. Therefore this study is to investigate the correlation and agreement between the intraocular pressure peaks detected during the water drinking test and modified diurnal tension curve in glaucomatous eyes and to analyze whether this is associated with prognostic outcome. The study will also measure autonomic nervous system activation during the test to investigate one possible mechanism behind it. The primary measure is peak Intraocular pressure measurements from two different measures. Secondary measures include OCT angiography, postural blood pressure, heart rate, pupil diameter. Current and future rates of progression using visual field and optical coherence tomography (OCT) measures. This is a prospective method comparison study, of 40 primary open angle and normal tension glaucoma patients who will attend for a single visit. Inclusion criteria include those

* Able to give informed consent to participate in the study
* Aged between 18 and 80 years of age
* Clear optical media
* Spherical equivalent +-10 Dioptres
* Normal tension glaucoma proven by visual field testing or OCT imaging combined with clinical assessment.
* Primary open angle glaucoma proven by visual field testing or OCT imaging combined with clinical assessment

Following completion of the study, participants will be followed up in their usual clinic as part of their regular care. The participants' follow-up data which is routinely generated as part of the glaucoma care pathway will be accessed for 18 months following completion of participation with a view of correlating initial results with possible disease progression and other related outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed consent to participate in the study
* Aged between 18 and 80 years of age
* Clear optical media
* Spherical equivalent +-10 Dioptres
* Normal tension glaucoma proven by visual field testing or OCT imaging combined with clinical assessment.
* Primary open angle glaucoma proven by visual field testing or OCT imaging combined with clinical assessment.

Exclusion Criteria:

* Are using ocular hypotensive therapy, or have done so in the last 30 days
* Have any other known ocular disease (except glaucoma)
* Have serious cardiac or kidney disease (WDT contra-indication)
* Have swallowing difficulties associated with either a neurological or gastrointestinal condition.
* Patients with any contra-indication of drinking large amounts of water in a small period of time e.g. swallowing impairment, oesophageal stricture, gastric banding.
* Have secondary or narrow/closed angle glaucoma
* Patients submitted to any surgical procedure or laser intervention during the evaluation period

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary open-angle and normal tension glaucoma patients
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2021-03-17 (Actual); Primary Completion 2021-06-09 (Actual); Study Completion 2021-06-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Cordeiro, Study Chair — Imperial College Healthcare NHS Trust
Locations (1):
- Imperial College Ophthalmic Research Group, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yap TE, Gao Y, Ahmad H, Susanna F, Susanna R, Normando EM, Bloom PA, Cordeiro MF. Comparison of intraocular pressure profiles during the water drinking test and the modified diurnal tension curve. Eye (Lond). 2024 Jun;38(8):1567-1574. doi: 10.1038/s41433-024-02954-0. Epub 2024 Mar 7. PMID 38454171

RESULTS

PARTICIPANT FLOW:
Groups:
- Glaucoma Patients: Those included in the study were male or female participants between the ages of 18 to 80 years old with a diagnosis of POAG or NTG in either eye.
Period: Overall Study
Arm/Group | Glaucoma Patients
Started | 46
Completed | 42
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Glaucoma Patients
Number analyzed (Participants) | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.5 (9.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 42
Mean baseline IOP (± SD) [Mean (Standard Deviation); unit: mmHg] — IOP (intraocular pressure)
  mmHg | 14.9 (4.5)
Mean visual field mean deviation [Mean (Standard Deviation); unit: dB] — Measurement of the light intensity used to test (Decibels) Normally the more negative this number is the more severe is the condition.
  dB | -5.05 (5.45)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Intraocular Pressure Difference (Between mDCT and WDT)
Description: Maximum intraocular pressure difference between two methods applied to each subject (modified diurnal tension curve mDTC and water drinking test WDT). The difference between maximum intraocular pressure of five eye pressure measurements taken at 8:00, 10:00, 12:00, 14:00 and 16:00 minus the maximum intraocular pressure measured at 15 minute intervals over 45 minutes during the water drinking test.
Time Frame: Single measurement (mDCT 5 measurements taken one every 2 hours and WDT a measurement taken every 15 minutes up to 45 minutes)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Glaucoma Patients
Number analyzed (Participants) | 42
mmHg | -0.82 (2.06)

ADVERSE EVENTS:
Time Frame: 2.5 months
Arm/Group | Glaucoma Patients
All-Cause Mortality (participants affected / at risk) | 0/42
Serious Adverse Events (participants affected / at risk) | 0/42
Other Adverse Events (participants affected / at risk) | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-09-14): https://cdn.clinicaltrials.gov/large-docs/31/NCT05283031/Prot_SAP_ICF_000.pdf